CLINICAL TRIAL: NCT05807438
Title: Comparison of the Immediate Effects of Physiotherapist and Self-administered Myofascial Release Techniques on Flexibility and Jumping Ability in Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YEDITEPEU-BUSRAKOCAKILIC-00096
Record Dates: First submitted 2023-03-16; First posted 2023-04-11 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Myofascial Spasm
MeSH Terms: interventions — Myofascial Release Therapy; Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The statistician and the physiotherapist who performed the tests were blinded to the study, and the participants were also blinded to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Foam Roller group (Active Comparator): Myofascial release with foam roller, hamstring and gastrocnemius muscle groups were trained with foam roller for 30 seconds with 2 repetitions
  Interventions: Other: Self myofascial Release
- Manual myofascial release group(Hands on) (Active Comparator): We used the following treatment protocol for all patients in the MFR group. The techniques were performed by a physiotherapist with experience in MFR.
  Interventions: Other: myofascial release

INTERVENTIONS:
Other: Self myofascial Release — Myofascial release participants on their own will roll the foam roller in each area for two minutes.
  Other Names: SMFR
  Arms: Foam Roller group
Other: myofascial release — Myofascial release will be applied to the participants by the physiotherapist.
  Other Names: Hands-on
  Arms: Manual myofascial release group(Hands on)

SUMMARY:
Basketball is an aerobic-based anaerobic sport that calls for both high-intensity movements like jumping (for rebounds, blocks, and shots), spins, dribbling, sprinting, and screening and low-intensity movements like walking, stopping, and running.This sport requires sudden and fast movements where jumping performance is often a decisive factor for sporting success and Whether crouching in a defensive situation or throwing a long pass, a player needs to have a sufficient level of flexibility for adequate efficiency. Fascia connects the structures of the body with muscles, nerves and blood vessels. Limitations may occur due to injury. These limitations can reduce flexibility, strength, endurance and coordination.Therefore, this study aims to compare the acute effects of manual and self-myofascial release on flexibility and jump performance in basketball players. The secondary aim was to examine the acute improvements in flexibility and jump performance after myofascial therapy.

DETAILED DESCRIPTION:
Basketball is a sport that changes very fast and quickly on the court and involves being always ready and mobile to pass, shoot, dribble or rebound. Some performance-related physical fitness parameters of basketball are: speed, flexibility, endurance, body composition, strength, agility, coordination. Some performance-related physical fitness parameters of basketball are: speed, flexibility, endurance, body composition, strength, agility, coordination.As a result of the high thrust forces generated during jumping and the eccentric forces applied to the lower body during landing, these athletes place great stress on their ankles and knees and require a high degree of force application and the ability to safely control eccentric landing forces.These functional changes are mainly controlled by the lower limbs, but lower limb control is influenced by range of motion, which affects flexibility when strength is reduced." It is easy to see why flexibility is so important for effective basketball sport efficiency.Flexibility is important in both prevention and rehabilitation of musculoskeletal injuries. When looking at sports performance, the hamstring and gastrocnemius muscles have a fundamental role in the myofascial chain defined by Myers. Myofascial release is a series of manual therapy techniques that involve applying pressure to soft tissue (fascia) to achieve structural and mechanical adaptation.The therapist applies a continuous, slow and steady pressure on the restricted tissue barrier and when the tissue relaxes, a new tissue barrier is applied.While continuous pressure applied to fascia tissue is called direct treatment and traction applied is called indirect treatment, another treatment method is self-myofascial release. Self-Myofascial Release (SMR) is performed by applying pressure on restricted fascia tissue using various materials and one's own body weight in different body positions. The material used can be foam roller, vibrating foam roller.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 45 years of age,
* gastrocnemius and hamstring muscle injuries. absence of pes planus and plantar heel pain

Exclusion Criteria:

* presence of a disease in which manual application cannot be performed (tumour, fracture, rheumatoid arthritis, osteoporosis, severe vascular disease, etc.),
* history of surgery in the lower extremity in the last 6 months,
* diagnosis of fibromyalgia syndrome,
* chronic pain

Ages: 15 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-08 (Estimated); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-05-04 (Estimated)

PRIMARY OUTCOMES:
counter movement jump(CMJ) | a day before the rehabilitation
  Players were asked to jump as high as possible; the highest jump will then was recorded in centimeter scoring: The timing mat may give a score of the time in the air, and the calculated vertical jump height can be calculated. Height can be calculated using this formula: jump height = 4.9 x (0.5 x Time)^2 ). The jump height is usually greater than achieved with the Squat Jump.
counter movement jump(CMJ) | at the time of discharge(2 weeks)
  Players were asked to jump as high as possible; the highest jump will then was recorded in centimeter scoring: The timing mat may give a score of the time in the air, and the calculated vertical jump height can be calculated. Height can be calculated using this formula: jump height = 4.9 x (0.5 x Time)^2 ). The jump height is usually greater than achieved with the Squat Jump.
Squat jump (SJ) | a day before the rehabilitation
  The squat jump test measures explosive strength. This test is performed by starting with your knees bent in a 90 degree angle, and jumping vertically as high as possible from that position. Hands should be held on the hips to avoid the effect of arm swinging to the test.
Squat jump (SJ) | at the time of discharge(2 weeks)
  The squat jump test measures explosive strength. This test is performed by starting with your knees bent in a 90 degree angle, and jumping vertically as high as possible from that position. Hands should be held on the hips to avoid the effect of arm swinging to the test.

SECONDARY OUTCOMES:
sit and reach test | a day before the rehabilitation
  The sit and reach test will be used to assess lumbar and hamstring flexibility will be applied. The sit and reach test will be performed through the lumbopelvic region and hamstrings It is widely used to estimate flexibility. Sit with your feet in a V shape touching the tape, feet about a foot apart, with the measuring tape in between your legs, the 0 end starting where your legs part. Overlap your hands with arms outstretched in front of you. Practice three times, leaning forward and reaching your hands out.
sit and reach test | at the time of discharge(2 weeks)
  The sit and reach test will be used to assess lumbar and hamstring flexibility will be applied. The sit and reach test will be performed through the lumbopelvic region and hamstrings It is widely used to estimate flexibility. Sit with your feet in a V shape touching the tape, feet about a foot apart, with the measuring tape in between your legs, the 0 end starting where your legs part. Overlap your hands with arms outstretched in front of you. Practice three times, leaning forward and reaching your hands out.
knee - wall tests | a day before the rehabilitation
  The test requires a wall and a measuring tape. The measuring tape is attached to the wall touching and placed on the floor perpendicular to the wall. Tape the participant's foot is asked to step on it. The heel and 2nd toe are asked to be on the line. The participant then tries to touch the knee to the vertical line drawn on the wall ahead. The participant can use support while moving forwards. The participant should place his/her foot on the line. takes the knee as far as it can go without lifting it. In the last case, the test at the moment when the knee of the leg touches the wall and the heel of the foot on the tape touches the floor the measurement will take place at the point where it will be pressed. To understand the test and to ensure that the correct measurement.3 measurements will be made in order to be taken. The big toe of the foot tested with the wall distance (cm) will be noted. The best of three trials for data analysis will be taken into account.
knee - wall tests | at the time of discharge(2 weeks)
  The test requires a wall and a measuring tape. The measuring tape is attached to the wall touching and placed on the floor perpendicular to the wall. Tape the participant's foot is asked to step on it. The heel and 2nd toe are asked to be on the line. The participant then tries to touch the knee to the vertical line drawn on the wall ahead. The participant can use support while moving forwards. The participant should place his/her foot on the line. takes the knee as far as it can go without lifting it. In the last case, the test at the moment when the knee of the leg touches the wall and the heel of the foot on the tape touches the floor the measurement will take place at the point where it will be pressed. To understand the test and to ensure that the correct measurement.3 measurements will be made in order to be taken. The big toe of the foot tested with the wall distance (cm) will be noted. The best of three trials for data analysis will be taken into account.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Tuğçe Çil, doctor, Study Director — Yeditepe University
Locations (3):
- Turkey (Türkiye) (3):
  - Elif Tuğçe, Istanbul, Maltepe
  - Hazal, Istanbul, Maltepe
  - Büşra, Istanbul, Maltepe

IPD SHARING:
Plan to Share IPD: No